CLINICAL TRIAL: NCT06134271
Title: A Multicenter, Prospective, Cohort Study on the Treatment of Metastatic Hormone-sensitive Prostate Cancer Patients Who Have Progressed After Pre-treatment With Rezvilutamide Combined With Abiraterone
Brief Title: Rezvilutamide Plus Abiraterone for Metastatic Hormone-sensitive Prostate Cancer
Acronym: RASTOM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jianbin Bi (Other)
Responsible Party: Sponsor-Investigator, Jianbin Bi, Director of Urology Department, the First Hospital of China Medical University, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstHCMU-JBi-RASTOM
Record Dates: First submitted 2023-10-29; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
Keywords: prostate cancer; rezvilutamide; abiraterone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rezvilutamide cohort (Experimental): Rezvilutamide 240 mg orally once a day. Patients should also receive androgen deprivation therapy, which includes both gonadotropin releasing hormone analogue (GnRHa) castration treatment or bilateral orchiectomy.
  Interventions: Drug: Rezvilutamide
- Rezvilutamide plus abiraterone cohort (Experimental): Rezvilutamide 240 mg orally once a day. Simultaneously, take orally 1000 mg of Abiraterone tablets and 5 mg of prednisone once a day. Patients should also receive androgen deprivation therapy simultaneously, that is, they should also receive gonadotropin releasing hormone analogue (GnRHa) castration treatment or have undergone bilateral orchiectomy.
  Interventions: Drug: Rezvilutamide plus abiraterone
- Continue previous treatment cohort (Experimental): Continue using the previous treatment regimen for treatment.
  Interventions: Drug: Continue previous treatment

INTERVENTIONS:
Drug: Rezvilutamide — Rezvilutamide 240mg qd
  Arms: Rezvilutamide cohort
Drug: Rezvilutamide plus abiraterone — Rezvilutamide 240mg qd plus abiraterone 1000mg + prednisone 5 mg qd
  Arms: Rezvilutamide plus abiraterone cohort
Drug: Continue previous treatment — Continue using the previous treatment regimen for treatment.
  Arms: Continue previous treatment cohort

SUMMARY:
This multicenter, prospective, cohort study enrolled patients with metastatic hormone-sensitive prostate cancer who had been treated with other novel endocrine or systemic regimens (excluding patients treated with pre-order chemotherapy alone or bicalutamide); To observe the efficacy and safety of rezvilutamide alone or in combination with abiraterone in hormone-sensitive prostate cancer patients with PSA progression following prior sequence therapy.

DETAILED DESCRIPTION:
This is a multicenter, prospective, cohort study to observe the efficacy and safety of rezvilutamide alone or in combination with abiraterone in patients with hormone-sensitive prostate cancer who have progressed PSA after prior sequencing therapy. Other novel endocrine or systemic regimens were used in these patients (excluding patients treated with pre-order chemotherapy alone or bicalutamide); and received ongoing gonadotropin-releasing hormone analogue (GnRHa) castration therapy (drug castration) or prior bilateral orchiectomy (surgical castration) over the course of the study; Participants who did not undergo bilateral orchiectomy had to maintain effective pharmacological castration throughout the study period.

This study included three cohorts of 160 patients with progressive metastatic hormone-sensitive prostate cancer. 56 patients were included in cohort 1, 56 patients in cohort 2 and 28 patients in cohort 3. Patients in cohort 1 were treated with rezvilutamide, 240 mg/day; Patients in cohort 2 received rezvilutamide at 240 mg/day in combination with abiraterone and hormonal therapy; Patients in cohort 3 maintained promiscuous therapy until disease progression or uncontrolled toxicity. According to PCWG3, the primary endpoint is Time to CRPC. Secondary endpoints included OS, rPFS, time to SEE, liver function assessment, and safety of NCI-TCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; male;
2. Patients with pathological detection of prostate cancer and clinical diagnosis of metastatic hormone-sensitive patients with bone scanning, electronic computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET-CT) and other imaging examinations;
3. Patients with mHSPC are allowed to use other novel endocrine or systemic regimens in the pre-order (excluding those treated with chemotherapy alone or bicalutamide), castration with an ongoing gonadotropin-releasing hormone analogue (GnRHa) (drug castration), or prior bilateral orchiectomy (surgical castration); Participants who did not undergo bilateral orchiectomy had to maintain effective pharmacological castration throughout the study period;
4. PSA progression at enrollment: for patients who respond to initial therapy, PSA progression is determined if serum PSA exceeds 25% of the minimum PSA during treatment and > 0.4 ng/mL in absolute terms, and after repeated confirmation 3 weeks after the elevation is found; for patients with persistent PSA elevation after initial treatment, PSA progression is determined when the PSA elevation exceeds 25% of the baseline value and the absolute value is>0.4 ng/mL at 12 weeks of treatment;
5. The Eastern Cooperative Oncology Group（ECOG）PS of 0 or1;
6. The main organ indicators such as blood routine, coagulation function, liver and kidney function, and heart function are normal:

   * ANC≥1.5×109/L；
   * PLT≥100×109/L
   * Hb≥90g/L；
   * TBIL≤1.5×ULN；
   * ALT and AST≤2.5×ULN；
   * BUN（or UREC）和Cr≤1.5×ULN；
   * LVEF≥50%； Volunteer to participate in this clinical trial, understand the research procedure, and have signed an informed consent form

Exclusion Criteria:

1. Failure to sign an informed consent form;
2. Patients with allergic reactions to the pharmaceutical ingredients or excipients used in the study;
3. Patients with difficulty swallowing or poor digestion and absorption function；
4. Patients with severe liver function impairment (Child Pugh C grade)；
5. Confirmed by imaging, there is a brain tumor lesion; Having a history of epilepsy, or having a disease that can trigger seizures within the 12 months prior to C1D1 (including a history of transient ischemic attacks, stroke, traumatic brain injury with consciousness disorders requiring hospitalization);
6. Active heart disease within the first 6 months of C1D1, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and ventricular arrhythmias requiring medication;
7. Suffering from any other malignant tumor within the first 5 years of C1D1 (excluding fully remitted in situ cancer and malignant tumors that have been determined by the researchers to progress slowly);
8. Have a history of immunodeficiency (including HIV testing positive, other acquired or congenital immunodeficiency diseases) or a history of organ transplantation;
9. Subjects who are unwilling to take effective contraceptive measures during the entire study treatment period and within 30 days after the last administration;
10. According to the judgment of the investigator, there are concomitant diseases (such as poorly controlled hypertension, serious diabetes, neurological or mental diseases, etc.) or any other conditions that seriously endanger the safety of patients, may confuse the research results, or affect the completion of the study by the subjects;
11. Patients participating in other clinical trial studies; After evaluation by the researcher, any other circumstances deemed unsuitable for participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to castration-resistant prostate cancer (CRPC) | From the first day of patient enrollment until the time reach CRPC, the duration of the assessment should not exceed 24 months.
  The time reach CRPC is defined as the occurrence of the following events, whichever occurs first, serum PSA progression: PSA value>2 ng/ml, interval of 1 week, consecutive 2 times, increase>50% from baseline, serum testosterone at castrated level (<50 ng/dL or 1.7 nmol/L) or soft tissue, visceral imaging progression or bone injury (following the recommendations of Prostate Cancer Clinical Trial Working Group 3 [PCWG3]); Imaging progression of soft tissue/visceral lesions based on magnetic resonance imaging (MRI)/computed tomography (CT) performed by researchers on the chest, abdomen, and pelvis (based on RECIST 1.1).

SECONDARY OUTCOMES:
Overall survival (OS) | From the first day of patient enrollment to all-cause mortality, the duration of the assessment should not exceed 24 months.
  Overall survival is defined as the time from the first day of enrollment to the patient's death due to any cause.
Radiographic Progression-free survival (rPFS) | From the first day of patient enrollment to the time reach radiographic progression, the duration of the assessment should not exceed 24 months.
  The radiographic progression free survival is defined as the time from the first day of patient enrollment to imaging progression or death. Imaging progress includes progress under bone scanning, where at least 2 new lesions are discovered under bone scanning, or measurable soft tissue lesions are detected under computed tomography (CT) or magnetic resonance imaging (MRI) (based on the definition of the Solid Tumor Response Evaluation Standard (RECIST) version 1.1). According to RECIST 1.1 guidelines, progression requires a 20% increase in the sum of all target lesion diameters, and an absolute minimum sum increase of 5 millimeters (mm) compared to the sum of the lowest values.
Time to first Symptomatic Skeletal Event (SSE) | From the first day of patient enrollment to the occurrence of the SSE, the duration of the assessment should not exceed 24 months.
  Symptomatic Skeletal Event (SSE) is defined as the occurrence of the following events, including fractures, spinal cord compression, bone specific radiotherapy or surgery, and death from any cause, whichever occurs first.radiotherapy or surgery for bones, death for all cause, whichever occurs first.
Liver function assessment | From the first day of patient enrollment to the end of treatment, the evaluation duration should not exceed 24 months
  Liver function will be assessed once every 2 weeks in the first three cycles, once every 4 weeks in the continues treatment.
Safety profile | From the first day of patient enrollment to the end of treatment, the evaluation duration should not exceed 24 months
  Any adverse events were recorded starting from the first administration of riviramide or the combination of riviramide and abiolone until the end of the safety follow-up period.Among them, liver function assessment is conducted in the first 3 cycles, once every 2 weeks; Subsequent treatment should be conducted once every 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbin Bi, Study Director — First Hospital of China Medical University

IPD SHARING:
Plan to Share IPD: No